CLINICAL TRIAL: NCT04843280
Title: Comparison of Traditional Physical Therapy to Internet-Based Physical Therapy After Knee Arthroscopy: A Prospective Randomized Controlled Trial Comparing Patient Outcomes and Satisfaction
Brief Title: Traditional PT v Internet Based PT After Total Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DMAZ17D.288
Record Dates: First submitted 2021-03-31; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Physical Therapy
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Physical Therapy (Active Comparator): Participants who have undergone primary unilateral knee arthroscopy will undergo 6 weeks of formal outpatient physical therapy
  Interventions: Procedure: Traditional Outpatient Physical Therapy
- Internet Based Physical Therapy (Active Comparator): Participants who have undergone primary unilateral knee arthroscopy will undergo 6 weeks of internet based rehabilitation regime in the home through the online recovery program, FORCE Therapeutics
  Interventions: Procedure: FORCE therapeutics (physical therapy)

INTERVENTIONS:
Procedure: FORCE therapeutics (physical therapy) — 6 weeks of internet based physical therapy following arthroscopic knee surgery
  Arms: Internet Based Physical Therapy
Procedure: Traditional Outpatient Physical Therapy — 6 weeks of outpatient physical therapy following arthroscopic knee surgery
  Arms: Traditional Physical Therapy

SUMMARY:
Knee arthroscopy results in significant improvements in functional outcomes, pain relief and quality of life for patients suffering from mechanical symptoms associated with meniscal tears. Patients are able to return to their activities of daily living, occupation, or sport without significant limitations. Traditionally, patients have undergone formal physical therapy (PT) after knee arthroscopy to regain function. There is a significant cost and time commitment associated with traditional outpatient physical therapy. An internet based therapy program allows patients to perform therapy at home on their own time schedule. A recent study demonstrated that patients who undergo internet based PT after total knee arthroplasty performed as well patients receiving traditional physical therapy. These findings have not been studied in the knee arthroscopy patient population. The goal of this study is to compare traditional outpatient physical therapy rehabilitation to Internet-based rehabilitation in patients undergoing knee arthroscopy for partial meniscectomy.

The purpose of this study is to compare functional outcome, and patient satisfaction, internet-based rehabilitation program vs. standard outpatient physical therapy after unilateral knee arthroscopy for meniscal tear.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing unilateral primary knee arthroscopy for meniscal tear
* Any patient 18 years or older

Exclusion Criteria:

* Patients without access to the Internet
* Post-traumatic osteoarthritis
* Patients with ligamentous injury
* Patients with full thickness cartilage defects
* Patients with osteoarthritis or inflammatory arthritis
* Revision or conversion knee arthroscopy
* Patients receiving workers compensations
* Patients discharged to a rehabilitation unit or other form of respite care such as a skilled nursing facility, acute rehabilitation center, convalescent home, long-term care facility or nursing home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2017-07-30 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Postoperative Knee Function | 4 months
  Investigators will be measuring whether there is an increase in participants function as assessed by the International Knee Documentation Committee (IKDC) Subjective Knee Evaluation. This will be measured on a scale of 0-100 with 0 being the lowest level of function and 100 being the highest level of function
Cost analysis | 4 months
  cost analysis survey will be completed by participants to determine if there is a difference in outpatient physical therapy versus internet based physical therapy
Postoperative Physical therapy Patient Satisfaction | 4 months
  Participant satisfaction with physical therapy will be assessed using the physical therapy satisfaction evaluation. This consist of a single question asking the participant how satisfied they are with their surgery on a scale of 0-10. 0 being not satisfied at all and 10 being extremely satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States